CLINICAL TRIAL: NCT06743867
Title: A Prospective, Multi-center, Single-arm Clinical Research Evaluating the Safety and Efficacy of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) for Peritoneal Metastatic Adenocarcinoma
Brief Title: The Safety and Efficacy of Pressurized Intraperitoneal Aerosol Chemotherapy for Peritoneal Metastatic Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Tianjin Third Central Hospital (Other); Peking University Cancer Hospital & Institute (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Henan Cancer Hospital (Other Government); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Jiangxi Provincial Cancer Hospital (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Nanfang Hospital, Southern Medical University (Other); Southern Medical University, China (Other); Affiliated Hospital of Qinghai University (Other); Ruijin Hospital (Other); Shenzhen Second People's Hospital (Other); West China Hospital (Other); Tianjin Nankai Hospital (Other); Wannan Medical College Yijishan Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Changzhi People's Hospital (Other); First Hospital of China Medical University (Other); Xiangya Hospital of Central South University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Sun Yat-sen University (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC-HOPE-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Peritoneal Carcinoma Metastatic
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) (Experimental): Drug: Pressurized Intraperitoneal Aerosol Chemotherapy
  Interventions: Drug: Pressurized Intraperitoneal Aerosol Chemotherapy

INTERVENTIONS:
Drug: Pressurized Intraperitoneal Aerosol Chemotherapy — The comprehensive therapeutic strategy will be modified based on the integrated 2- or 3-week systemic chemotherapies. In the interim, a total of three PIPAC procedures will be conducted for all qualifying patients.
  1. PIPAC combined with 2-week systemic chemotherapies:
     PIPAC therapy will occur every four weeks, while systemic chemotherapies will be administered during the first and third weeks following the initial and second PIPAC procedures respectively.
  2. PIPAC combined with 3-week systemic chemotherapies:
  (1) Scheme 1: PIPAC therapy will occur every 6 weeks, with systemic chemotherapies administered during the 1st and 4th weeks following the first and second PIPAC procedures, respectively.
  (2) Scheme 2: PIPAC therapy will occur every 6 weeks, while systemic chemotherapies will be administered in the 2nd and 5th weeks following the initial and second PIPAC procedures, respectively.
  Other Names: Systemic chemotherapy

SUMMARY:
This research is a prospective, multi-center, single-arm clinical trial aimed at assessing the standard pressurized intraperitoneal aerosol chemotherapy (PIPAC) utilizing a novel nebulized drug delivery system (NDDS) for patients with peritoneal metastatic adenocarcinoma (PMA) originating from gastric, colorectal, appendiceal, or ovarian cancer.

The primary objectives of this study are to assess the safety and efficacy of PIPAC with the novel NDDS in the treatment of PMA. Primary endpoints include adverse events (AEs) and serious AEs, as assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, incidences of device defects, postoperative pain scores evaluated using the Visual Analogue Scale / Score (VAS), and quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 scale, Version 3.0). Secondary endpoints include the intra-abdominal peritoneal cancer index (PCI), peritoneal regression grading score (PRGS), objective response rate (including partial response (PR) and complete response (CR)), improvement in ascites, conversion rate (patients proceeding to cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) following initial PIPAC treatments), progression-free survival (PFS), and overall survival (OS).

DETAILED DESCRIPTION:
Peritoneal metastasis (PM) is acknowledged as the final stage of various abdominal cancers and correlates with dismal prognosis, with survival generally under six months when exclusively managed with systemic chemotherapy due to the plasma-peritoneal barrier. Recent clinical evidence, primarily from Western nations, has shown that pressurized intraperitoneal aerosol chemotherapy (PIPAC) is a viable, safe, and effective method for PM. Nonetheless, clinical data regarding the utilization of PIPAC in Asian populations, especially among Chinese patients, are still scarce. This study seeks to evaluate the safety and efficacy of PIPAC employing a novel nebulized drug delivery system (NDDS) for the treatment of peritoneal metastatic adenocarcinoma (PMA).

The NDDS novel consists of a central computer with an operating system, a high-pressure peristaltic pump, an emergency stops switch, a liquid level sensor, and an integrated unit featuring a 10-mm spray nozzle, an anti-high-pressure infusion tube, and a puncture head. PIPAC is conducted under a standard 12 mmHg pneumoperitoneum. Doxorubicin and cisplatin are administered for patients with PMA originating from gastric or ovarian cancers, whereas oxaliplatin is utilized for PMA resulting from colorectal or appendiceal cancers. Customized treatment protocols, encompassing drug dosages, are established by a multidisciplinary peritoneal carcinomatosis committee before the administration of PIPAC.

Qualified patients will undergo three cycles of PIPAC in conjunction with concurrent systemic chemotherapy (e.g., XELOX or FOLFOX). The interval between successive PIPAC procedures is 4 to 6 weeks, with an additional interval of one to two weeks between PIPAC and systemic chemotherapy. The anticipated therapy duration for each patient is three months, during which the primary and secondary endpoints will be assessed.

This research will take place in 25 domestic medical centers, aiming for a sample size of 30 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology verified that peritoneal metastatic adenocarcinoma (PMA) arises from gastric, colorectal, appendiceal, or ovarian carcinoma;
2. Applicable to individuals of either sex, aged between 18 and 75 years;
3. Eastern Cooperative Oncology Group (ECOG) scale ≤ 2;
4. Absence of other concurrent malignancies;
5. Without contraindications for laparoscopic surgery;
6. Laboratory testing: blood routine examination: neutrophil count ≥ 1.5× 10^9/L, platelet count ≥ 80 × 10^9/L, hemoglobin ≥ 80g/L ; blood biochemistry: serum total bilirubin ≤ 1.5 ×ULN, Alanine transaminase and aspartate aminotransferase ≤ 2.5 ×ULN, serum creatinine ≤ 1.5 ×ULN;
7. Life expectancy > 6 months;
8. Informed consent understood and signed.

Exclusion Criteria:

1. Presenting symptoms of gastrointestinal obstruction;
2. Fully reliant on parenteral nutrition;
3. Exhibiting decompensated ascites;
4. Suffering from severe abdominal infection (indications of peritonitis);
5. Characterized by extensive adhesions in the abdominal cavity;
6. Concurrently undergoing cytoreductive surgery (CRS) or gastrointestinal tract resection and reconstruction procedures;
7. With portal vein thrombosis;
8. Concurrently, individuals with significant or unmanaged medical conditions or infections (including atrial fibrillation, angina, cardiac dysfunction, ejection fraction < 50%, refractory hypertension etc.);
9. Previous chemotherapeutic drugs allergy;
10. Severe cardiopulmonary, hepatonephric, hematologic, and metal diseases, or drug abuse;
11. Pregnancy or lactating women;
12. Engage in additional clinical trials within three months preceding recruitment;
13. Other conditions: patients are inappropriately included as determined by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) and serious AE associated with Treatment | 4-6 weeks following the initial and secondary PIPAC procedures, and 6 months subsequent to the tertiary PIPAC procedure
  Treatment-related adverse events are categorized according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Elevated grades correlate with increased severity of adverse events
Incidences of device defects | During each PIPAC therapy
  Incidences of device defects during PIPAC therapy
Postoperative pain scores | The first to seventh day after the PIPAC procedure
  Postoperative pain is assessed using the Visual Analogue Scale/Score (VAS), which integrates the Wong-Baker Faces Pain Scale Revision (FPS-R) and the Numerical Rating Scale (NRS). Scores vary from 0 to 10, with 1-3 indicating "mild pain (sleep unaffected)", 4-6 indicating "moderate pain (sleep disruption)", and 7-10 indicating "severe pain (severe sleep disruption)".
Quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Version 3.0) | 4-6 weeks following the initial and second PIPAC procedures, and 6 months subsequent to the third PIPAC procedure
  The quality of life is assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 scale, Version 3.0). A higher comprehensive score indicates superior quality of life.

SECONDARY OUTCOMES:
Intra-abdominal peritoneal cancer index (PCI) | During each PIPAC procedure
  The peritoneal cancer index (PCI) is assessed based on the presence and dimensions of peritoneal metastases in various areas of the abdominal cavity. Elevated PCI scores indicate a greater peritoneal tumor burden.
Peritoneal regression grading score (PRGS) | During each PIPAC procedure
  The peritoneal regression grading score is assessed through the pathological examination of biopsies from the four quadrants (right upper/lower and left upper/lower) of the anterior abdominal wall, correlating with the ratio of residual active to necrotic tumor cells. The grading scores span from 1 to 4, with lower scores indicating fewer residual active tumor cells.
Objective response rate (partial and complete response) | Within 6 months after the third PIPAC procedure
  The objective response rate, encompassing both partial and complete responses, is assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Improvement in ascites | During each PIPAC procedure
  The volume and hue of ascites are documented and assessed
Conversion rate | 4-6 weeks following the initial and secondary PIPAC procedures, and 6 months after the tertiary PIPAC procedure
  The conversion rate is defined as the percentage of PMA patients who could subsequently undergo cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) following initial PIPAC treatments in this study
Progression-free survival (PFS) | 6 months after the second or third PIPAC procedure
  Duration from the commencement of PIPAC treatment to the advancement of the disease
Overall survival (OS) | 6 months after the second or third PIPAC procedure
  Duration from the commencement of PIPAC treatment to mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China